CLINICAL TRIAL: NCT03153969
Title: A Clinical Trial to Evaluate a New Giomer Restorative System in Class V Restorations
Brief Title: Clinical Evaluation of a New Giomer Restorative System in Class V Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Shofu Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Gerard Kugel, Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12486
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Non-carious Cervical Lesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SHOFU Beautifil II LS (Experimental): Composite: SHOFU Beautifil II LS, Bonding Agent: SHOFU BeautiBond
  Interventions: Device: SHOFU Beautifil II LS
- 3M/ESPE Filtek Supreme (Active Comparator): Composite: 3M/ESPE Filtek Supreme, Bonding Agent: 3M/ESPE Scotchbond Universal
  Interventions: Device: 3M/ESPE Filtek Supreme

INTERVENTIONS:
Device: SHOFU Beautifil II LS — Placed under manufacturer's instructions
  Arms: SHOFU Beautifil II LS
Device: 3M/ESPE Filtek Supreme — Placed under manufacturer's instructions
  Arms: 3M/ESPE Filtek Supreme

SUMMARY:
The objective of this study is to evaluate the clinical effectiveness of a new composite resin (SHOFU Beautifil II LS) vs a control (3M/ESPE Filtek Supreme) for use in restoring non carious cervical lesions Class V lesions.

3M ESPE FiltekTM Supreme is one of the composite resin materials that will be used in this study (Group 1). This is a light-activated, flowable restorative composite.

Shofu Beautifil II LS (SI R21204) is a new type of filling material called a Giomer. This is the second composite that will be used in this study (Group 2) Giomer is a collective term for dental materials that will release ions, such as fluoride. Results from previous studies show that the released ions may have beneficial effects on the tooth, including strengthening the tooth.

In each participant, one tooth with a class V lesion will be randomized to group 1, and a second tooth with a class V lesion will be randomized to group 2. The restorations will be observed over 18 months to determine clinical acceptability.

DETAILED DESCRIPTION:
This is a single-center, non-blinded, controlled, split mouth, clinical trial 18 months in duration.

The purpose of this clinical trial is to evaluate the effectiveness of a new Giomer restorative system (Shofu Beautifil LS) for use in restoring non carious Class V lesions by comparing it to 3M ESPE FiltekTM Supreme in the following categories:

Clinical Assessments (Documentation at baseline, 6months and 18months):

* Surface Luster
* Surface Staining
* Marginal Staining
* Color Match
* Anatomical Form
* Marginal Adaptation
* Fracture of Material and Retention
* Radiographic Examination
* Patient's View
* Postoperative Hypersensitivity
* Recurrence of Caries
* Tooth Integrity
* Adjacent Mucosa

Sensitivity interview- assessed preoperatively (prior to anesthesia, if needed) at baseline and after restoration placement

Dentin Sclerosis Rating- assessed at baseline

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, in general health
* Must have a minimum of 2 cervical lesions in need of restoration
* Cervical lesions must provide for a minimum of 1mm thickness of restorative material while maintaining natural tooth contour
* At least 50% of lesion must be in dentin
* Coronal margin of lesion must be in enamel

Exclusion Criteria:

* Rampant uncontrolled caries
* Systemic or local disorders that contra-indicate the dental procedures included in this study
* Evidence of xerostomia
* Evidence of severe bruxing or clenching or in need of TMJ related therapy
* Women who are pregnant or breast feeding (self-reported).
* Known allergy to resin composites or local anesthetics
* Abnormal oral soft tissue findings (e.g., open sores, lesions)
* Condition affecting salivary flow (e.g., salivary gland disorder, Sjögren's Syndrome)
* Teeth with periapical pathology or exhibiting symptoms of pulpal pathology
* Teeth that are non-vital or have had root canal therapy
* Teeth that have been pulp capped
* Teeth with near exposures on pre-operative radiographs
* Hypersensitive teeth
* Teeth with a periodontal pocket of more than 4mm with bleeding on probing
* Teeth that are used as abutments for removable partial dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Hickel Criteria | Up to 18 months
  Clinical assessments (Esthetic properties: surface luster, surface staining, marginal staining, color match, anatomical form, Functional properties: marginal adaptation, fracture of material and retention, radiographic examination, patient's view, and Biological Properties: postoperative hypersensitivity, recurrence of caries, tooth integrity and adjacent mucosa) will be performed by two trained examiners other than the operating clinician using modified Hickel criteria at baseline and follow-up visits. Differences between the two groups for Hickel criteria items will be examined with the Wilcoxon signed-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Kugel, DMD, MS, PhD, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No